CLINICAL TRIAL: NCT05427604
Title: To Evaluate the Effects of Omega 3 Fatty Acids in the Context of Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Omegaserum
Record Dates: First submitted 2022-05-30; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential intervention (Other): 1. single ingestion of olive oil for assessement of monounsaturated fatty acids peak time in blood (3g)
  2. single ingestion of olive oil for collection of blood sample at peak time (3g)
  3. single ingestion of DHA-rich oil for assessement of polyunsaturated fatty acids peak time in blood (3g)
  4. single ingestion of DHA-rich oil for collection of blood sample at peak time (3g)
  Interventions: Other: Olive oil; Other: DHA oil

INTERVENTIONS:
Other: Olive oil — ingestion of olive oil (3g) and blood measurement at baseline, after 1h, 2h, 3h, 4h, 5h, 6h
Other: Olive Oil — ingestion of olive oil (3g) and blood sampling at the fatty acids pic concentration (for in vitro study)
Other: DHA oil — ingestion of DHA oil (3g) and blood measurement at baseline, after 1h, 2h, 3h, 4h, 5h, 6h
Other: DHA oil — ingestion of DHA oil (3g) and blood sampling at the fatty acids pic concentration (for in vitro study)

SUMMARY:
Previous studies have demonstrated, in an in vitro micro-tumour model (the spheroid) and in a mouse model, that long-chain omega-3 fatty acids, in particular docosahexaenoic acid (DHA), can inhibit tumour development.

Therefore, the aim of this study was to collect DHA-enriched human serum, following ingestion of a DHA-enriched oil, in order to assess its effect on tumour development in vitro. Blood enriched in fatty acids not containing DHA will be used as a control condition, obtained after ingestion of olive oil.

This study is an important step to determine the interest of DHA supplementation as a new approach to prevent tumour development, and/or as an adjuvant to cancer treatments.

DETAILED DESCRIPTION:
The objective of this study is to collect DHA-enriched human serum in order to test it on the in vitro tumour model, spheroids. The results will be compared with human serum enriched in fatty acids (saturated, monounsaturated and polyunsaturated) but not in DHA.

To do this, the study will be divided into 4 steps

1. determination of the time when a maximum concentration of fatty acids is observed in the serum after ingestion of olive oil (the control condition)
2. blood sampling at baseline (fasting) and at Tmax after olive oil ingestion
3. determination of the time when a maximum concentration of fatty acids is observed in the serum after ingestion of DHA-enriched oil (the test condition)
4. blood sampling at baseline (fasting) and at Tmax after ingestion of DHA-enriched oil.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 65 years;
* Body mass index between 20 and 30 kg/m2;
* For women: use of effective contraception;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Uncontrolled systolic blood pressure > 160/100 mmHg;
* For premenopausal women: pregnant women or women planning to get pregnant within 3 months or lactating women;
* For menopausal women: less than 6 months of menopause;
* Type II diabetes (controlled or uncontrolled), Type I diabetes;
* Medical history or actual severe psychiatric, severe neurologic, severe hepatic, severe pancreatic, severe kidney, severe pulmonary, severe cardiovascular or severe gastrointestinal problem;
* Thyroid disorder;
* Cancer < 3 years before the inclusion;
* Consumption of drug under prescription or over-the-counter drug or dietary supplement (including n-3 PUFA) within 1 month before the inclusion (excepted contraception);
* Consumption of fish or of omega-3 enriched eggs > 2 times per week within 1 month before the inclusion;
* Subjects who are not able to understand and follow study procedures;
* Drug addiction problem (occasional or regular consumption);
* Women who drink more than 2 glasses of alcohol per day (> 20 g of alcohol per day or > 140 g/week) or men who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day or more than 210 g/week);
* Subjects having given their blood within less than 3 months before inclusion;
* Subjects having participated to another clinical trial with an investigational product within less than 1 month before the inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Palmitoleic fatty acid pattern | through study completion, an average of 4 months
  Area under the curve of palmitoleic fatty acid in serum calculated during 6 hours post-ingestion
Docosahexaenoic fatty acid pattern | through study completion, an average of 4 months
  Area under the curve of docosahexaenoic acid in serum calculated during 6 hours post-ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain - CICN, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No